CLINICAL TRIAL: NCT01276418
Title: ENT FiberLase CO2 Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lumenis Be Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LUM-SBUSUR-ACF-09-01
Record Dates: First submitted 2011-01-09; First posted 2011-01-13 (Estimated); Last update posted 2016-09-07 (Estimated); Status verified 2012-01

CONDITIONS: Laryngeal Diseases; Pharyngeal Diseases
MeSH Terms: conditions — Laryngeal Diseases; Pharyngeal Diseases | interventions — Lasers, Gas

ARMS (1):
- Treatment (Experimental)
  Interventions: Device: CO2 laser

INTERVENTIONS:
Device: CO2 laser — Ablation and coagulation of soft tissue
  Other Names: Acupulse WG CO2 Laser; Fiberlase Flexible Fiber

SUMMARY:
This study is intended to collect data regarding treatment with a new flexible fiber used to transmit laser emitted from a Carbon dioxide (CO2) laser to the transoral region. This study will include a single treatment that is performed transorally (through the mouth) for oral or laryngeal indications in the field of Ear, Nose and Throate (ENT).

ELIGIBILITY:
Inclusion Criteria:

1. General good health allowing patient to undergo general anaesthesia or heavy sedation according to the specific procedure.
2. Adult
3. Able and willing to comply with all visit, treatment and evaluation schedule and requirements
4. Able to understand and provide written Informed Consent
5. Disease which requires tissue ablation for treatment

Exclusion Criteria:

1. Having a bleeding disorder or taking anticoagulation medications, including heavy use of aspirin, in a manner which does not allow for a minimum 10 day washout period prior to each treatment (as per the patient's physician discretion);
2. Significant concurrent illness, such as uncontrolled diabetes i.e. any disease state that in the opinion of the Physician would interfere with the anesthesia, treatment, or healing process
3. Mentally incompetent, prisoner or evidence of active substance or alcohol abuse;
4. Any condition which, in the Physician's opinion, would make it unsafe (for the subject or for the study personnel) to treat the subject as part of this research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2010-10; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Ability to complete procedure with the study device | Immediate - during intervention
  The number of interventions that were completed using the AcuPulse WG and FiberLase CO2 Fiber for the intended indication, without the need to revert to other means
Complications (bleeding, perforation, damage to non target tissue) | During intervention and up to 6 weeks following the procedure
  Number of subjects with Adverse Events as a Measure of Safety

CONTACTS AND LOCATIONS:
Locations (2):
- University Hospital of Mont-Godinne, Yvoir, Belgium
- Bufalini Hospital, Cesena, Italy